CLINICAL TRIAL: NCT00063934
Title: A Phase 1/2 Study of Bcl-2 Antisense Oligonucleotide G3139 in Combination With Doxorubicin and Docetaxel in Metastatic and Locally Advanced Breast Cancer
Brief Title: Oblimersen Plus Doxorubicin and Docetaxel in Treating Patients With Metastatic or Locally Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02885; NCI-2012-02885 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6023; DM02-700 (Other: M D Anderson Cancer Center); 6023 (Other: CTEP); P30CA016672 (NIH); N01CM17003 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Male Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — oblimersen; Doxorubicin; Docetaxel; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim

ARMS (1):
- Treatment (oblimersen, doxorubicin, docetaxel) (Experimental): PHASE I (COMPLETED AS OF 8/16/04): Patients receive oblimersen IV continuously on days 1-6 interrupted only to administer doxorubicin IV over 15 minutes and docetaxel IV over 60 minutes on day 6. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 7-13 or pegfilgrastim SC on day 7. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  PHASE II: Patients receive doxorubicin, docetaxel, G-CSF or pegfilgrastim, and oblimersen at the MTD as in phase I.
  Patients with resectable tumors after 6 courses undergo surgical resection.
  Interventions: Biological: oblimersen sodium; Drug: doxorubicin hydrochloride; Drug: docetaxel; Biological: filgrastim; Biological: pegfilgrastim; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF
Procedure: therapeutic conventional surgery — Undergo surgical resection
Other: pharmacological study — Optional correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of oblimersen when given together with doxorubicin and docetaxel and to see how well they work in treating women with metastatic or locally advanced breast cancer. Drugs used in chemotherapy, such as doxorubicin and docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of doxorubicin and docetaxel by making the tumor cells more sensitive to the drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the pharmacokinetics of G3139, doxorubicin and docetaxel in breast cancer patients receiving G3139/AT therapy. (Phase I) II. To determine the safety of bcl-2 antisense oligonucleotide G3139 (GenasenseTM) together with docetaxel plus doxorubicin (AT) in patients with metastatic and locally advanced breast cancer (LABC). (Phase I) III. To determine the therapeutic efficacy of neoadjuvant G3139 in combination with AT chemotherapy in patients with LABC. (Phase II) IV. To further evaluate the safety of bcl-2 antisense oligonucleotide G3139 (GenasenseTM) together with docetaxel plus doxorubicin (AT) in patients with locally advanced breast cancer (LABC). (Phase II)

SECONDARY OBJECTIVES:

I. To determine the clinical and imaging response to neoadjuvant G3139/AT in the breast and the axillary lymph nodes. (Phase II) II. To determine the disease-free survival of breast cancer patients treated with neoadjuvant G3139/AT. (Phase II) III. To further define the pharmacokinetics of G3139/AT. (Phase II) IV. To evaluate the role of Bcl-2 expression as a predictor of response to neoadjuvant G3139/AT therapy. (Phase II) V. To obtain serial breast cancer samples from patients treated with G3139. (Phase II)

OUTLINE: This is an open-label, dose-escalation study of oblimersen.

PHASE I (COMPLETED AS OF 8/16/04): Patients receive oblimersen IV continuously on days 1-6 interrupted only to administer doxorubicin IV over 15 minutes and docetaxel IV over 60 minutes on day 6. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 7-13 or pegfilgrastim SC on day 7. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive doxorubicin, docetaxel, G-CSF or pegfilgrastim, and oblimersen at the MTD as in phase I.

Patients with resectable tumors after 6 courses undergo surgical resection.

Patients are followed every 3-6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Patients must have histologically or cytologically confirmed breast cancer
* PHASE I: To be eligible for the phase I component of this study, patients must have stage IIIB, IIIC or IV breast cancer; these include patients with T4, any N, M0; any T, N3, M0; any T, any N, M1
* PHASE I: Measurable disease is not required for patients participating in the phase I component
* PHASE I: Prior G3139, taxane or anthracycline therapy is not allowed
* PHASE I: Patients may have received up to 3 prior chemotherapy regimens for breast cancer (excluding anthracyclines and taxanes), either as adjuvant/neoadjuvant therapy or for metastatic disease
* PHASE I: Life expectancy of greater than 6 months
* PHASE I: ECOG performance status =< 2 (Karnofsky >= 60%)
* PHASE I: Leukocytes >= 3,000/L
* PHASE I: Absolute neutrophil count >= 1,500/L
* PHASE I: Platelets >= 100,000/L
* PHASE I: Total bilirubin =< 1.5 mg/dl
* PHASE I: ALT(SGPT) =< 2.5 X upper limit of normal
* PHASE I: Creatinine =< 2.0 mg/dl
* PHASE I: Normal cardiac function (LVEF >= 45%) as documented by MUGA scan and/or echocardiogram
* PHASE I: The effects of G3139 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because anthracycline and taxanes used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* PHASE I: Ability to understand and the willingness to sign a written informed consent document
* PHASE II: Patients must have histologically or cytologically confirmed breast cancer
* PHASE II: Patients must have stage IIIA, IIIB, or IIIC breast cancer; these include patients with T4, any N, M0; any T, N2-3, M0; T3, N1, M0; patients with ipsilateral supraclavicular lymph node metastases (IIIC) are eligible; patients with evidence of distant metastases (stage IV) are not eligible
* PHASE II: Measurable disease is required; disease will be measured prior to initiation of G3139/doxorubicin/docetaxel therapy by physical exam, mammography and ultrasound of the affected areas; pathologic response will be measured at the time of definitive surgery
* PHASE II: Prior G3139 therapy is not allowed
* PHASE II: Prior chemotherapy, hormone therapy, definitive surgery, or radiation therapy for breast cancer are not allowed
* PHASE II: Life expectancy of greater than 6 months
* PHASE II: ECOG performance status =< 2 (Karnofsky >= 60%)
* PHASE II: Leukocytes >= 3,000/L
* PHASE II: Absolute neutrophil count >= 1,500/L
* PHASE II: Platelets >= 100,000/L
* PHASE II: Total bilirubin =< 1.5 mg/dl
* PHASE II: ALT(SGPT) =< 2.5 X upper limit of normal
* PHASE II: Creatinine =< 2.0 mg/dl
* PHASE II: Normal cardiac function (LVEF >= 45%) as documented by MUGA scan and/or echocardiogram
* PHASE II: The effects of G3139 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because anthracycline and taxanes used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* PHASE II: Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* PHASE I: Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the phase I study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* PHASE I: Patients may not be receiving any other investigational agents
* PHASE I: Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* PHASE I: Leptomeningeal disease
* PHASE I: Symptomatic lymphangitic pulmonary metastases
* PHASE I: History of allergic reactions attributed to compounds of similar chemical or biologic composition to G3139 or other agents used in the study; patients are excluded if known hypersensitivity to drugs formulated in polysorbate 80 (Tween 80)
* PHASE I: Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* PHASE I: Patients with neuropathy grade 2 or higher
* PHASE I: Pregnant women are excluded from this study because G3139 is an oligonucleotide agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with G3139, breastfeeding should be discontinued if the mother is treated with G3139; these potential risks may also apply to other agents used in this study, such as doxorubicin and docetaxel
* PHASE II: Patients may not be receiving any other investigational agents
* PHASE II: History of allergic reactions attributed to compounds of similar chemical or biologic composition to G3139 or other agents used in the study; patients are excluded if known hypersensitivity to drugs formulated in polysorbate 80 (Tween 80)
* PHASE II: Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* PHASE II: Patients with neuropathy grade 2 or higher
* PHASE II: Pregnant women are excluded from this study because G3139 is an oligonucleotide agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with G3139, breastfeeding should be discontinued if the mother is treated with G3139; these potential risks may also apply to other agents used in this study, such as doxorubicin and docetaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Esteva, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 16, 2003 to August 25, 2005; All recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 31 participants enrolled, one participant was ineligible for treatment.
Groups:
- Oblimersen Plus Doxorubicin + Docetaxel: Intravenous Oblimersen 7 mg/kg/day, both Doxorubicin 50 mg/m^2 and Docetaxel 75 mg/m^2 infused on Day 6
Period: Overall Study
Arm/Group | Oblimersen Plus Doxorubicin + Docetaxel
Started | 31
Completed | 30
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Groups:
- Neoadjuvant G3139, Doxorubicin and Docetaxel: Patients with locally advanced breast cancer received intravenous G3139 in combination with doxorubicin and docetaxel . Cycles were repeated every 21 days x 6.
Arm/Group | Neoadjuvant G3139, Doxorubicin and Docetaxel
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 49 [24 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Toxicities
Time Frame: From baseline until the date of first documented toxicity or date of death from any cause, whichever came first, assessed every three weeks up to 2 years and 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Oblimersen Plus Doxorubicin + Docetaxel
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR)
Description: Pathologic complete responses (pCR), defined as no evidence of residual invasive tumor, including no residual tumor in the axillary lymph nodes, measured by microscopic evaluation of tissue specimen at time of definitive surgery (after 6 courses of neoadjuvant therapy). Neoadjuvant (preoperative) therapy administered on the first five days of every 3-week cycle. Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000]
Time Frame: At time of definitive surgery (after 6 courses of neoadjuvant therapy in 3 week cycles), approximately 18 weeks
Population: Intention to treat eligible participants per protocol.
Measure: Number; unit: Participants
Arm/Group | Oblimersen Plus Doxorubicin + Docetaxel
Number analyzed (Participants) | 30
Participants | 0

3. Secondary Outcome: Clinical Imaging Responses
Description: Evaluation target lesions (clinical response) by physical exam/ultrasound measurements of primary tumor and axillary lymph nodes after 3-6 courses: Complete Response: Disappearance of all target lesions; Partial Response: >30% decrease in sum longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease: >20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of 1>new lesions; Stable Disease: Neither sufficient shrinkage for PR nor increase for PD, reference smallest sum LD since treatment started.
Time Frame: After 3 and 6 courses of 21 day treatments (up to 18 weeks)
Measure: Number; unit: participants
Arm/Group | Oblimersen Plus Doxorubicin + Docetaxel
Number analyzed (Participants) | 30
participants
  CR | 30
  PR | 0

4. Secondary Outcome: Bcl-2 Expression in Breast Cancer Tissue
Description: Number of participant with Bcl-2 Expression in breast cancer tissue by protein and mRNA expression before treatment and at 3-5 days after oblimersen treatment.
Time Frame: before treatment and at 3-5 days after oblimersen treatment
Measure: Number; unit: participants
Arm/Group | Oblimersen Plus Doxorubicin + Docetaxel
Number analyzed (Participants) | 30
participants | 30

ADVERSE EVENTS:
Time Frame: 2 years and 5 months
Arm/Group | Oblimersen Plus Doxorubicin + Docetaxel
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 30/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oblimersen Plus Doxorubicin + Docetaxel (N=30)
Infection, non-neutropenia (Infections and infestations) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Metabolism and nutrition disorders) | 4 (4)
Infection or fever with Neutropenia (Infections and infestations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (Endocrine disorders) | 21 (21)
Death (Cardiac disorders) | 1 (1) — The cause of death was most likely acute heart failure secondary to cardiomegaly and hypertension, complicated by severe acute diverticulitis.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oblimersen Plus Doxorubicin + Docetaxel (N=30)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Drug fever (General disorders) | 11 (11)
Fatigue (General disorders) | 9 (9)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 28 (28)
Ocular/Vision (other) (Eye disorders) | 2 (2)
Pruritis/Itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 6 (6)
Sensory Neuropathy (Nervous system disorders) | 3 (3) — Neurolgy
Stomatitis (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 12 (12)
Alanine aminotransferase (Hepatobiliary disorders) | 8 (8)
Neutropenia (Infections and infestations) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 21 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less